CLINICAL TRIAL: NCT03751852
Title: Body-Mind-Spirit Intervention for Women With Early Psychosis: a Randomized Controlled Trial
Brief Title: Body-Mind-Spirit Intervention for Women With Early Psychosis
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: The University of Hong Kong (Other)
Responsible Party: Principal Investigator, Professor Eric Y.H. Chen, Chi-li Pao Foundation Professor of Psychiatry; Chair Professor in Psychiatry; Head, Department of Psychiatry, The University of Hong Kong
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: JCWowExercise; 124-01 (Other: KWC IRB / REC No.)
Record Dates: First submitted 2018-06-14; First posted 2018-11-23 (Actual); Last update posted 2021-04-14 (Actual); Status verified 2021-04

CONDITIONS: Psychosis
MeSH Terms: conditions — Psychotic Disorders

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Exercise coaching group (Experimental): This intervention is an integration of aerobic exercise, yoga, mindfulness and exercise coaching. Exercise class and coaching will be provided weekly in the first 8 weeks. In the next 8 week, exercise class will be provided weekly while exercise coaching will be provided bi-weekly. The exercise class includes aerobic exercise coached by a well-trained intervention officer, and the yoga and mindfulness coached by a certified yoga instructor. The exercise coaching session followed by some stretching and aerobic exercise session. Both motivational coaching and aerobic exercise will be coached by a well-trained intervention officer.
  Interventions: Behavioral: Exercise Coaching
- Psychoeducation group (Active Comparator): This group is similar with the exercise coaching group while exercise coaching session will be substituted by psychoeducation session.
  Interventions: Behavioral: Psychoeducation

INTERVENTIONS:
Behavioral: Exercise Coaching — 28 classes in 16 weeks
  Arms: Exercise coaching group
Behavioral: Psychoeducation — 28 classes in 16 weeks
  Arms: Psychoeducation group

SUMMARY:
This is an open-labelled randomised controlled trial (RCT) that aims to examine the effectiveness of exercise coaching approach in improving the physical activity engagement in patients with psychosis.

DETAILED DESCRIPTION:
Patients with psychosis will be recruited from the out-patient department (OPD) of the Kwai Chung Hospital (KCH). The patient with informed consent will be randomly assigned to exercise coaching or psychoeducation group to prevent decline in cognitive and functional outcomes known to be common in this group. This comprises locally-tested evidence-based intervention strategies such as exercise and Yoga intervention, combined with exercise coaching to consolidate the exercise habit. Each of the intervention includes 28 sessions spanning for16-week.

ELIGIBILITY:
Inclusion Criteria:

* Female
* Age from 18-64
* Based on the Fifth version of the Diagnostic and Statistical Manual of Mental Disorders diagnosis to have schizophrenia and related psychotic disorders
* Have the ability to understand Chinese
* Able to give informed consent
* Physically fit for participating in our study assessed by using the Physical Activity Readiness Questionnaire (PAR-Q)

Exclusion Criteria:

* Severe physical illness (Myocardial Infarction, Hypertension, Fracture, Spinal problems in which exercise may be contraindicated), and seizure disorders.
* Comorbid substance dependence
* Unstable psychotic symptoms
* Any history of brain trauma or organic brain disease
* Known history of intellectual disability or special school attendance
* Other mental conditions that requires other treatment priorities, e.g., suicidal risk.
* Other medical conditions that severely limits participation, comprehension, or adherence to the treatment or assessment e.g., epilepsy, dementia, terminal medical illness.

Ages: 18 Years to 64 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Gender Based: Yes — As agreement with funder
Enrollment: 57 (Estimated)
Dates: Start 2018-11-15 (Actual); Primary Completion 2021-06-30 (Estimated); Study Completion 2021-09-30 (Estimated)

PRIMARY OUTCOMES:
Physical Activity Engagement | Change from baseline to 6-month post-intervention
  Measured by the Chinese Version of International Physical Activity Questionnaire (IPAQ-C)

CONTACTS AND LOCATIONS:
Overall Officials: Eric Yu Hai Chen, MD, Principal Investigator — The University of Hong Kong
Locations (1):
- University of Hong Kong, Hong Kong, Hong Kong

IPD SHARING:
Plan to Share IPD: No